CLINICAL TRIAL: NCT04464070
Title: Novel Pathways of Eicosanoid Metabolism
Brief Title: Pathways of Eicosanoid Metabolism
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Claus Schneider, Associate Professor of Pharmacology, Vanderbilt University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 150895
Record Dates: First submitted 2020-07-01; First posted 2020-07-09 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Metabolism of Prostaglandin D2
MeSH Terms: interventions — Niacin; Aspirin; Prostaglandin D2

STUDY DESIGN:
Intervention Model Description: Participants may be participating in all 4 arms of the study or in less than 4 arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- niacin (Experimental): Blood (10 ml) will be drawn from the subject. Immediately before or after the blood draw the subject will collect a urine (3-10 ml) sample. After the baseline blood draw and the urine sample is collected the subject will take 500 mg of niacin. The niacin will not be an extended release formulation. Subjects will be encouraged to drink plenty of water during the study. Subjects are instructed to collect urine 1, 2, 4, 6, 8, and 10 hours after niacin administration. Subjects will collect their urine in separate plastic tubes that will be provided to them.
  Approximately 1-2 h after niacin administration a second blood sample (10 ml) will be drawn from the subject.
  Interventions: Dietary Supplement: niacin
- niacin + low-dose aspirin (Experimental): Volunteers will provide a urine sample. They will receive 7 tablets of low-dose aspirin (81 mg) and be instructed to take one tablet daily for 7 days. On the seventh day, they return to have blood drawn, urine collected, and receive niacin as described in arm 1.
  Interventions: Dietary Supplement: niacin; Drug: aspirin
- niacin + regular-strength aspirin (Experimental): Volunteers will provide a urine sample. They will receive 7 tablets of regular-strength aspirin (325 mg) and be instructed to take one tablet daily for 7 days. On the seventh day, they return to have blood drawn, urine collected, and receive niacin as described in arm 1.
  Interventions: Dietary Supplement: niacin; Drug: aspirin
- deuterated PGD2 (Experimental): Volunteers will come to the clinical research center. Volunteers will provide a urine sample. The volunteers will be fitted to record an electrocardiogram (ECG) and blood pressure. ECG will be recorded continuously. Blood pressure will be taken at baseline and every 10 minutes thereafter for one hour. The solution with deuterated PGD2 (10 microgram) will be infused over the course of 30 min. Volunteers will be monitored for 1 h after the end of the infusion, and volunteers will start collecting urine in intervals up to 10 h.
  Infusion of the deuterated PGD2 solution will be performed in the presence of a physician. The injection solution will be prepared by Vanderbilt University Medical Center (VUMC) Investigational Drug Services. The solution will be sterile and pyrogen free.
  Interventions: Other: PGD2

INTERVENTIONS:
Dietary Supplement: niacin — induce biosynthesis of PGD2
  Arms: niacin; niacin + low-dose aspirin; niacin + regular-strength aspirin
Drug: aspirin — inhibition of cyclooxygenase
  Arms: niacin + low-dose aspirin; niacin + regular-strength aspirin
Other: PGD2 — labeled precursor
  Arms: deuterated PGD2

SUMMARY:
Prostaglandins are important signaling compounds formed from arachidonic acid. The enzymes that form prostaglandins, cyclooxygenase-1 and -2 are the targets of non-steroidal anti-inflammatory drugs (NSAIDs). Because prostaglandins are very unstable in the body, they can not be measured directly. Instead, their metabolites are isolated from urine or blood and quantified as markers of formation of the parent, active compounds.

The investigators are testing the hypothesis that there is a previously unrecognized metabolic pathway between two prostaglandins. The investigators hypothesize that prostaglandin D2 (PGD2), in addition to its known metabolism to PGD-M, is also metabolized to 11-dehydro-thromboxane B2 (11-dehydro-TxB2).

DETAILED DESCRIPTION:
The objective of this study is to determine whether PGD2 is metabolized to 11-dehydro-TxB2 in humans. Because the levels of PGD2 and its metabolite, PGD-M, are low in human urine, the investigators will use the model of niacin-induced flushing which is associated with a increased release of PGD2 from skin cells. It has been demonstrated that increased formation of PGD2 is associated with increased levels of urinary 11-dehydro-TxB2 in patients with mastocytosis.

In order to test whether niacin-induced biosynthesis of PGD2 is associated with formation of 11-dehydro-TxB2 the investigators will measure prostaglandin metabolites in blood and urine of volunteers receiving niacin. In addition, subjects will be treated with low or high dose aspirin prior to niacin to analyze the contribution of cyclooxygenase enzymes to biosynthesis of PGD2.

Arm 1: Subjects will receive 500 mg niacin. The subjects will collect urine (3-10 ml each) before niacin and every one-two hours after niacin for 10 h. Subjects will have blood drawn (2 teaspoons) before and at 0.5-1 h after niacin.

Arm 2: Subjects will take 81 mg aspirin (1 tablet of low-dose aspirin) daily for 7 days before niacin. Urine collection will be before and after aspirin, before niacin, and then in intervals as in arm 1. There will be a blood collection before niacin and 0.5-1 h after niacin.

Arm 3: Subjects will take 325 mg aspirin (1 tablet of regular strength aspirin) daily for 7 days before niacin. Urine collection will be before and after aspirin, before niacin, and then in intervals as in arm 1.

Arm 4: Subjects will be infused with 10 μg of deuterated PGD2 in a forearm vein over the course of 30 min. Subjects will collect a urine sample before and every two hours after deuterated PGD2 for 10 h.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy volunteers not currently taking any medication.

Exclusion Criteria:

* Use of anti-inflammatory/over-the-counter pain medications (NSAIDs) up to 2 weeks prior to study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-08-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
prostaglandin metabolites | 0-10 hours
  metabolites will be quantified in urine and blood

CONTACTS AND LOCATIONS:
Overall Officials: Claus M Schneider, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD (study protocol, informed consent forms) will be shared upon a justified request by an investigator.
Supporting Information: Study Protocol, ICF
Time Frame: IPD will become available from the beginning of the study until completion.
Access Criteria: Researchers need to make a justified request.